CLINICAL TRIAL: NCT06088095
Title: The Effect of Gradual Mobilization on Vital Signs and Comfort Level After Transfemoral Coronary Angiography
Brief Title: Comfort Level After Transfemoral Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Özlem Ceyhan, Director, TC Erciyes University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: coronary angiography
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-02

CONDITIONS: Coronary Disease
Keywords: comfort; coronary angiography; vital signs
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Mobility group
- control group (No Intervention)

INTERVENTIONS:
Other: Mobility group — Patients will be mobilized in accordance with the gradual mobilization procedure 12 hours after the angiography procedure.
  Arms: intervention group

SUMMARY:
With the increase in the number of cardiovascular diseases, the safety of the angiography method used in diagnosis and treatment becomes important. The transfemoral approach is often preferred during angiography. It is recommended to have bed rest for 6-12 hours after transfemoral angiography (TFA) to prevent possible complications. In order to reduce the complications arising from angiography, it is predicted from the studies that giving the patient a therapeutic position, elevating the head of the bed and gradual early mobilization will reduce the patients' groin pain, prevent urinary retention and increase patient comfort. In this study, the effect of gradual mobilization after transfemoral angiography on the vital signs, complications and comfort level of the patients. It is planned to be done to determine the

ELIGIBILITY:
Inclusion Criteria:

* Individuals who can be contacted at a level that can answer research questions
* Individuals with transfemoral angiography

Exclusion Criteria:

* Those with hypertension
* Individuals with psychological and neurological disorders
* Patients with communication problems
* Patients with deterioration in hemodynamics after angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Pulse rate per minute | 20 minutes
  Vital signs
blood pressure rate, mmHg | 20 minutes
  Vital signs
respiratory rate per minute | 20 minutes
  Vital signs
SpO2 value of the patients will be measured. | 20 minutes
  Vital signs

SECONDARY OUTCOMES:
General Comfort Scale | The comfort scale will be filled 2 hours after mobilization.
  It is used to determine the comfort level of patients. The highest score that can be given to the positive items in the scale, four (4), indicates high comfort, and the lowest score, one (1), indicates low comfort. Thus, the lowest score that can be obtained in the GAS is 48 points, while the highest score is 192 points. As the score obtained from the scale increases, the comfort level perceived by the patient increases. The total score obtained is divided by 48, which is the number of scale items, and the average value is found in the range of 1-4. If the patient performing the scale has low comfort, it is expressed as one (1), and if the patient has high comfort, it is expressed as four (4).

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsaman SEA. Association of position change and back massage and early ambulation with post-transfemoral coronary angiography complications. J Vasc Nurs. 2022 Sep;40(3):128-133. doi: 10.1016/j.jvn.2022.08.003. Epub 2022 Sep 11. PMID 36414367
- [Background] Ramos Dos Santos PM, Aquaroni Ricci N, Aparecida Bordignon Suster E, de Moraes Paisani D, Dias Chiavegato L. Effects of early mobilisation in patients after cardiac surgery: a systematic review. Physiotherapy. 2017 Mar;103(1):1-12. doi: 10.1016/j.physio.2016.08.003. Epub 2016 Sep 14. PMID 27931870
- [Background] Ibdah RK, Ta'an WF, Shatnawi RM, Suliman MM, Rababah JA, Rawashdeh SI. The effectiveness of early position change postcardiac catheterization on patient's outcomes: A randomized controlled trial. Nurs Forum. 2020 Jul;55(3):380-388. doi: 10.1111/nuf.12438. Epub 2020 Feb 5. PMID 32020631
- [Background] Rezaei-Adaryani M, Ahmadi F, Asghari-Jafarabadi M. The effect of changing position and early ambulation after cardiac catheterization on patients' outcomes: a single-blind randomized controlled trial. Int J Nurs Stud. 2009 Aug;46(8):1047-53. doi: 10.1016/j.ijnurstu.2009.02.004. Epub 2009 Mar 17. PMID 19296949